CLINICAL TRIAL: NCT03692130
Title: Mindfulness, Acceptance and Commitment Combined in Cognitive Behavioral Group Therapy (MAC-CBT®) for Patients With Depression
Brief Title: Treatment of Depression With Mindfulness, Acceptance and Commitment
Acronym: MAC_Depr
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neuropsychiatrischen Zentrums Hamburg-Altona (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Peter Tonn, Director, Neuropsychiatrischen Zentrums Hamburg-Altona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCHULZE02
Record Dates: First submitted 2018-08-23; First posted 2018-10-02 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Psychotherapy; Depression
Keywords: Acceptance; Mindfulness; Commitment; Group-Psychotherapy
MeSH Terms: conditions — Depression | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: One group with new treatment, one group with known and defined treatment
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants don't know in which of the both arms they are, the outcome assessor don't know which participant of which study-arm he/she calculate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Treatment (Active Comparator): The patients will be treated with psychological group treatment for 8 Sessions with focus on mindfulness, acceptance and commitment in a special adapted treatment process.This will be called "Mindfulness, Acceptance and Commitment-Therapy for depressive Patients".
  Interventions: Behavioral: Mindfulness, Acceptance and Commitment-Therapy
- Known Treatment (Sham Comparator): The participants will be treated with a relaxation-treatment, long time established as "jacobson muscle relaxing technique".
  Interventions: Behavioral: Jacobson

INTERVENTIONS:
Behavioral: Mindfulness, Acceptance and Commitment-Therapy — Psychotherapeutic intervention to treat depressive patients with special exercises and education to be mindful, to accept situations and behaviors and to commit with the situation or the possibility to change.
  Arms: New Treatment
Behavioral: Jacobson — Relaxation treatment in technique of Jacobson
  Arms: Known Treatment

SUMMARY:
Randomized trial to proof the effects and efficacy of a new mindfulness and acceptance based group-treatment for depressive patients

DETAILED DESCRIPTION:
In this study, a randomized trial is conducted in which the participants are allocated to two different care services (MAC-CBT® vs. progressive muscle relaxation). Participants are patients with depression who have been made aware of the group therapy by their treating physicians or psychotherapists or who have read the advertising in waiting areas or on the investigators homepage. An extensive psychometric survey will be conducted at the start of the study in an interview session with a psychotherapist, who also judges if the participants are able to participate in a therapy group. The MAC-CBT® group receives an eight-session group therapy, in which the aspects of mindfulness, acceptance and commitment are taught in detail. The control group will receive an eight-session treatment with progressive muscle relaxation. Input and output results are determined using validated survey instruments. In addition, the investigators will check the data for moderating variables (e.g. age, gender, previous treatments...).

ELIGIBILITY:
Inclusion Criteria:

* Depressive Disorder

Exclusion Criteria:

* Somatic disorder
* psychotic disorder
* personality disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Depression - Patient Health Questionnaire-9 | Measurement of PHQ-Data 3 months after inclusion of participant
  Measurement of changes of depressive Symptoms, so called PHQ-9. There will be a measure of the total score, range from 9 to 36, pathological in sense of depression will be any score above 15. There is only one measurement scale (PHQ-9) with nine items, no other measurements or different units in the PHQ-9.

SECONDARY OUTCOMES:
Quality of Life - European Quality 5 Dimensions on 3 Levels | Measurement of QoL 3 months after inclusion of participant
  Measurements of changes of Quality of life (EQ-5D 3L), there will be a measure of three dimensions of life quality in scores 0-10, the total is a sum and will be added from the single measurements. There is a range from 0-30, no "critical number" is defined, only the sum will be used for interpretation. A higher score represents a better result /state
Anxiety - Generalized Anxiety Disorder | Measurement of Generalized Anxiety 3 months after inclusion of participant
  Measurements of changes of Anxiety (GAD 7), there are 7 questions to check anxiety, the range is from 7-28, pathological in sense of manifest anxiety disorder is a sum above 9 plus the key-question.A lower score represents a better result/ state.
Acceptance and Commitment - Questionnaire of Mindfulness, Acceptance and Commitment (MAC-Q) | Measurement of Mindfulness, Acceptance and Commitment 3 months after inclusion of participant
  Measurements of changes of Mindfulness, Acceptance and Commitment, that is a measurement with 8 questions, range from 0-32, only the sum will be noticed, no "critics score" is published yet. A higher score represents a better result/ state.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tonn, MD, Principal Investigator — Managing Director
Locations (1):
- Neuropsychiatric Center of Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No